CLINICAL TRIAL: NCT00132730
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter, Parallel-Group, Dose-Ranging Study of MK-0873 in Patients With COPD
Brief Title: An Investigational Drug Study In Patients With COPD (Chronic Obstructive Pulmonary Disease) (MK-0873-005)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0873-005; 2005_015 (Other: Telerex Study ID)
Record Dates: First submitted 2005-08-03; First posted 2005-08-22 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Lung Diseases; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive | interventions — MK 0873

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- MK-0873 2.5 mg (Experimental): Participants receive placebo tablets once daily for 3 weeks in Period I (Base), MK-0873 2.5 mg tablets once daily for 12 weeks in Period II (Base) and MK-0873 2.5 mg tablets once daily for 12 weeks in Period III (EXT1)
  Interventions: Drug: MK-0873 2.5 mg; Drug: Placebo to MK-0873
- MK-0873 1.25 mg (Experimental): Participants receive placebo tablets once daily for 3 weeks in Period I (Base), MK-0873 1.25 mg tablets once daily for 12 weeks in Period II (Base) and MK-0873 2.5 mg tablets once daily for 12 weeks in Period III (EXT1)
  Interventions: Drug: MK-0873 1.25 mg; Drug: Placebo to MK-0873
- MK-0873 0.75 mg (Experimental): Participants receive placebo tablets once daily for 3 weeks in Period I (Base), MK-0873 0.75 mg tablets once daily for 12 weeks in Period II (Base) and MK-0873 2.5 mg tablets once daily for 12 weeks in Period III (EXT1)
  Interventions: Drug: MK-0873 0.75 mg; Drug: Placebo to MK-0873
- Placebo (Placebo Comparator): Participants receive placebo tablets once daily for 3 weeks in Period I (Base), placebo tablets once daily for 12 weeks in Period II (Base) and placebo tablets once daily for 12 weeks in Period III (EXT1)
  Interventions: Drug: Placebo to MK-0873
- MK-0873 2.5 mg + Usual Care (Experimental): Participants receive MK-0873 2.5 mg tablets once daily plus usual care (inhaled short- or long-acting beta-agonists, inhaled corticosteroids, or short- or long-acting anticholinergics) for 28 weeks during Periods IV and V (EXT2)
  Interventions: Drug: MK-0873 2.5 mg; Drug: Usual Care
- Usual Care (Active Comparator): Participants receive usual care (inhaled short- or long-acting beta-agonists, inhaled corticosteroids, or short- or long-acting anticholinergics) for 28 weeks during Periods IV and V (EXT2)
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: MK-0873 2.5 mg
  Arms: MK-0873 2.5 mg; MK-0873 2.5 mg + Usual Care
Drug: MK-0873 1.25 mg
  Arms: MK-0873 1.25 mg
Drug: MK-0873 0.75 mg
  Arms: MK-0873 0.75 mg
Drug: Placebo to MK-0873
  Arms: MK-0873 0.75 mg; MK-0873 1.25 mg; MK-0873 2.5 mg; Placebo
Drug: Usual Care
  Arms: MK-0873 2.5 mg + Usual Care; Usual Care

SUMMARY:
This is a study to evaluate the effectiveness and tolerability of a once-daily oral medication (MK-0873) for the treatment of COPD (chronic obstructive pulmonary disease) to determine whether the study drug leads to an improvement in pulmonary (lung) function, as well as symptoms, and quality of life.

DETAILED DESCRIPTION:
Following a three-week run-in period (Period I) during which participants received placebo, participants entered into a 12-week double-blind treatment period (Period II) during which they received daily doses of either one of three doses of MK-0873 or placebo. Period I and Period II made up the Base Study. Following the 12-week treatment period in the Base Study, participants were invited to continue in an optional 12-week double-blind extension study (Period III, EXT1). Participants who received any dose of MK-0873 in the Base Study continued on MK-0873 2.5 mg daily in Period III while participants in the placebo arm of the Base Study continued on placebo daily. Following EXT1, participants were invited to continue in an optional open-label second extension study (EXT2) which was to last 80 weeks (Period IV: 28 weeks, Period V: 52 weeks). In EXT2, participants who had been taking MK-0873 2.5 mg in the Base Study were allocated to MK-0873 2.5 mg plus usual care, while participants who had been taking the other two doses of MK-0873 or placebo in the Base Study were allocated to either MK-0873 2.5 mg plus usual care or to usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 40 to 75 years old, with a history consistent with COPD (chronic obstructive pulmonary disease)
* Lung function tests that meet the requirements of the study

Exclusion Criteria:

* Severe and unstable medical conditions other than COPD (chronic obstructive pulmonary disease)
* Use of continuous oxygen therapy
* Cardiac (heart) arrhythmias
* Other lung disease
* History of colitis (inflammation of the colon)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2004-06-01 (Actual); Primary Completion 2005-08-17 (Actual); Study Completion 2005-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0873-005&kw=0873-005&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0873 0.75 mg Base Study: Participants receive placebo tablets once daily for 3 weeks in Period I (Base), and MK-0873 0.75 mg tablets once daily for 12 weeks in Period II (Base)
- MK-0873 1.25 mg Base Study: Participants receive placebo tablets once daily for 3 weeks in Period I (Base), and MK-0873 1.25 mg tablets once daily for 12 weeks in Period II (Base)
- MK-0873 2.5 mg Base Study: Participants receive placebo tablets once daily for 3 weeks in Period I (Base), MK-0873 2.5 mg tablets once daily for 12 weeks in Period II (Base) and MK-0873 2.5 mg tablets once daily for 12 weeks in Period III (EXT1)
- Placebo Base Study: Participants receive placebo tablets once daily for 3 weeks in Period I (Base), placebo tablets once daily for 12 weeks in Period II (Base) and placebo tablets once daily for 12 weeks in Period III (EXT1)
- MK-0873 2.5 mg + Usual Care: Participants receive MK-0873 2.5 mg tablets once daily plus usual care (inhaled short- or long-acting beta-agonists, inhaled corticosteroids, or short- or long-acting anticholinergics) for 28 weeks in Periods IV and V (EXT2)
- Usual Care: Participants receive usual care (inhaled short- or long-acting beta-agonists, inhaled corticosteroids, or short- or long-acting anticholinergics) for 28 weeks in Periods IV and V (EXT2)
Period: Period I - Placebo Run-in (Base)
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study | MK-0873 2.5 mg + Usual Care | Usual Care
Started | 150 | 148 | 153 | 153 | 0 | 0
Completed | 150 | 148 | 153 | 153 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period II - 12-week Treatment (Base)
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study | MK-0873 2.5 mg + Usual Care | Usual Care
Started | 150 | 148 | 153 | 153 | 0 | 0
Completed | 127 | 133 | 135 | 131 | 0 | 0
Not Completed | 23 | 15 | 18 | 22 | 0 | 0
Not completed — Clinical adverse experience | 11 | 4 | 9 | 9 | 0 | 0
Not completed — Laboratory adverse experience | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Other reasons | 11 | 10 | 9 | 13 | 0 | 0
Period: Period III - Blinded Extension (EXT1)
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study | MK-0873 2.5 mg + Usual Care | Usual Care
Started | 0 | 0 | 317 (Includes all MK-0873 participants from Period II. Not all eligible participants entered EXT1) | 107 (Not all eligible participants entered EXT1) | 0 | 0
Completed | 0 | 0 | 235 | 82 | 0 | 0
Not Completed | 0 | 0 | 82 | 25 | 0 | 0
Not completed — Site terminated | 0 | 0 | 57 | 20 | 0 | 0
Not completed — Clinical adverse experience | 0 | 0 | 11 | 1 | 0 | 0
Not completed — Laboratory adverse experience | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other reasons | 0 | 0 | 14 | 3 | 0 | 0
Period: Period IV - Open-label Extension (EXT2)
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study | MK-0873 2.5 mg + Usual Care | Usual Care
Started | 0 | 0 | 0 | 0 | 187 (Includes participants from Period III. Not all eligible participants entered EXT2) | 71 (Includes paricipants from Period III. Not all eligible participants entered EXT2)
Completed | 0 | 0 | 0 | 0 | 8 | 3
Not Completed | 0 | 0 | 0 | 0 | 179 | 68
Not completed — Site terminated | 0 | 0 | 0 | 0 | 169 | 68
Not completed — Clinical adverse experience | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Laboratory adverse experience | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 6 | 0
Period: Period V - Open-label Extension (EXT2)
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study | MK-0873 2.5 mg + Usual Care | Usual Care
Started | 0 | 0 | 0 | 0 | 7 (Not all participants who completed Period IV entered Period V) | 2 (Not all participants who completed Period IV entered Period V)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 7 | 2
Not completed — Site terminated | 0 | 0 | 0 | 0 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- MK-0873 0.75 mg Base Study: Participants receive placebo tablets once daily for 3 weeks in Period I (Base), MK-0873 0.75 mg tablets once daily for 12 weeks in Period II (Base) and MK-0873 2.5 mg tablets once daily for 12 weeks in Period III (EXT1)
- MK-0873 1.25 mg Base Study: Participants receive placebo tablets once daily for 3 weeks in Period I (Base), MK-0873 1.25 mg tablets once daily for 12 weeks in Period II (Base) and MK-0873 2.5 mg tablets once daily for 12 weeks in Period III (EXT1)
- Total: Total of all reporting groups
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study | Total
Number analyzed (Participants) | 150 | 148 | 153 | 153 | 604
Age, Customized [Number; unit: participants] — Number of Participants Between 42 and 77 Years of Age
  participants | 150 | 148 | 153 | 153 | 604
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 45 | 45 | 41 | 167
  Male | 114 | 103 | 108 | 112 | 437

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pre-dose (Trough) Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is a measure, in liters, of the amount of air expired in 1 second. Measured values were averaged during the placebo run-in period for baseline and over the last 4 weeks of the 12-week treatment period for on-treatment. For participants who did not have any measurements over the last 4 weeks of the 12-week treatment period, the last available on-treatment measurement was carried forward.
Time Frame: Pre-dose at Baseline and Treatment Weeks 8, 10 and 12
Population: The modified intention-to-treat (ITT) population includes all participants who had a baseline and at least one posttreatment measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study
Number analyzed (Participants) | 147 | 143 | 153 | 152
liters | -0.005 [-0.032 to 0.023] | -0.037 [-0.065 to -0.009] | -0.015 [-0.043 to 0.012] | -0.010 [-0.038 to 0.017]

2. Secondary Outcome: Change From Baseline in Overall Daytime Symptoms Score
Description: On a daily diary card, participants rated their responses to the question "Overall, how much of the time did you have symptoms from your lung disease today?" (0=none of the time; 5=all of the time). Scores range from 0 to 5, with higher scores indicating more time with symptoms. The overall daytime symptoms score value was the mean daily diary score during the placebo run-in period for baseline and over the last 4 weeks of the 12-week treatment period for on-treatment.
Time Frame: Baseline and Treatment Weeks 8, 10 and 12
Population: The modified ITT population includes all participants who had a baseline and at least one posttreatment measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study
Number analyzed (Participants) | 145 | 144 | 149 | 148
score on a scale | -0.15 [-0.24 to -0.06] | -0.11 [-0.21 to -0.02] | -0.13 [-0.22 to -0.04] | -0.14 [-0.23 to -0.05]

3. Secondary Outcome: Change From Baseline in Total Daily Beta-agonist Use
Description: The total daily beta-agonist use was measured in puffs per day and was recorded on daily diary cards by participants. It is defined as the sum of beta-agonist use between when participants arose from and went to bed. The total daily beta-agonist use values were the recorded mean during the placebo run-in period for baseline and over the last 4 weeks of the 12-week treatment period for on-treatment.
Time Frame: Baseline and Treatment Weeks 8, 10 and 12
Population: The modified ITT population includes all participants who had a baseline and at least one posttreatment measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs per day of beta-agonist
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study
Number analyzed (Participants) | 141 | 140 | 146 | 145
Puffs per day of beta-agonist | -0.04 [-0.45 to 0.38] | -0.14 [-0.56 to 0.27] | 0.04 [-0.38 to 0.46] | 0.07 [-0.35 to 0.48]

4. Secondary Outcome: Change From Baseline in Saint George's Respiratory Questionnaire (SGRQ) Response
Description: The SGRQ consists of 76 items in 3 domains: Symptoms (frequency and severity), Activity (activities that cause or are limited by breathlessness) and Impacts (social functioning, psychological disturbances resulting from airways disease). Scores for each domain and a total score are calculated; each questionnaire response has a unique empirically dervied "weight". Scores range from 0 to 100, with higher scores indicating poor health. Each domain of the questionnaire is scored separately in 2 steps: 1) The weights for all items with a positive response are summed; 2) The score is calculated by dividing the summed weights by the maximum possible weight for that domain and expressing the results as a percentage. The mean SGRQ scores were calculated during the placebo run-in period for baseline and over the last 4 weeks of the 12-week treatment period for on-treatment.
Time Frame: Baseline and Treatment Weeks 8 and 12
Population: The modified ITT population includes all participants who had a baseline and at least one posttreatment measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study
Number analyzed (Participants) | 141 | 140 | 144 | 143
score on a scale | -2.92 [-4.69 to -1.16] | -3.26 [-5.03 to -1.49] | -2.08 [-3.85 to -0.31] | -3.22 [-4.99 to -1.46]

5. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score
Description: The baseline dyspnea index (BDI) was measured at the randomization visit as a 3-domain score with a scale of 0 to 4 in each domain, with a total focal score of 12 indicating no dyspnea limitation and 0 indicating severe dyspnea. After 12 weeks of treatment, the investigator-administered TDI was completed, with a change in each of the 3 domains being rated from -3 (major deterioration) to +3 (major improvement), so that the TDI focal score could range from -9 to +9. A higher TDI focal score indicates improvement.
Time Frame: Baseline and Treatment Week 12
Population: The modified ITT population includes all participants who had a baseline and at least one posttreatment measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study
Number analyzed (Participants) | 138 | 140 | 141 | 137
score on a scale | 1.41 (3.04) [0.95 to 1.88] | 1.49 (3.07) [1.03 to 1.94] | 1.41 (2.55) [0.95 to 1.87] | 1.66 (2.73) [1.20 to 2.12]

6. Secondary Outcome: Change From Baseline in Shortness of Breath Questionnaire (SOBQ) Response
Description: The SOBQ is a validated 24-item measure of dyspnea associated with activities of daily living in patients with moderate to severe chronic lung disease. Twenty-one items ask patients about how frequently they experience shortness of breath (SOB) on a 6-point scale of 0 (never) to 5 (activity given up due to dyspnea) when performing various tasks. Three additional questions about limitations due to SOB, fear of harm from overexertion and fear of SOB are included for a total of 24 items. If patients do not routinely perform the activity indicated in the questionnaire, they are asked to estimate the degree of SOB anticipated. The SOBQ total score is calculated by summing responses across all 24 items. The total score ranges from 0 to 120, with a higher score indicating greater frequency of and limitations due to SOB. The score assessed at the baseline visit was used for the baseline score and the mean score assessed at Treatment Weeks 8 and 12 was used as the on-treatment score.
Time Frame: Baseline and Treatment Weeks 8 and 12
Population: The modified ITT population includes all participants who had a baseline and at least one posttreatment measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study
Number analyzed (Participants) | 141 | 140 | 144 | 143
score on a scale | -2.90 [-5.06 to -0.74] | -3.12 [-5.29 to -0.96] | -2.28 [-4.44 to -0.12] | -1.08 [-3.24 to 1.07]

7. Secondary Outcome: Number of Participants With at Least One Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: COPD exacerbation is defined as any change in symptoms or functional status that leads to administration (at investigator's discretion) of systemic corticosteroids (above participant's usual dose) and/or antibiotics, or an unscheduled COPD-related hospitalization, emergency room visit, or doctor visit. The number of participants who experienced at least one COPD exacerbation during the 12-week treatment period is reported.
Time Frame: Baseline through Treatment Week 12
Population: The modified ITT population includes all participants who had a baseline and at least one posttreatment measurement.
Measure: Number; unit: participants
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study
Number analyzed (Participants) | 150 | 148 | 153 | 153
participants | 37 | 37 | 33 | 38

8. Secondary Outcome: Change From Baseline in Predose (Trough) Forced Vital Capacity (FVC)
Description: FVC is a measure, in liters and using a spirometer, of the amount of air forcibly exhaled from the lungs after taking the deepest breath possible. The values averaged during the placebo run-in period were used for the baseline measurement and the values averaged over Treatment Weeks 8, 10 and 12 were used for the on-treatment measurement. A higher value indicates greater lung exiratory function.
Time Frame: Predose at Baseline and Treatment Weeks 8, 10 and 12
Population: The modified ITT population includes all participants who had a baseline and at least one posttreatment measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study
Number analyzed (Participants) | 147 | 143 | 153 | 152
liters | 0.008 [-0.053 to 0.069] | -0.082 [-0.144 to -0.021] | -0.002 [-0.062 to 0.058] | -0.069 [-0.129 to -0.009]

ADVERSE EVENTS:
Time Frame: Up to 14 weeks in the Base Study; up to 14 weeks in study EXT1; up to 80 weeks in study EXT2
Groups:
- MK-0873 2.5 mg EXT 1: Participants receive MK-0873 2.5 mg tablets once daily for 12 weeks in Period III (EXT1)
- Placebo EXT 1: Participants receive placebo tablets once daily for 12 weeks in Period III (EXT1)
- MK-0873 2.5 mg + Usual Care EXT 2: Participants receive MK-0873 2.5 mg tablets once daily plus usual care (inhaled short- or long-acting beta-agonists, inhaled corticosteroids, or short- or long-acting anticholinergics) for 28 weeks in Periods IV and V (EXT2)
- Usual Care EXT2: Participants receive usual care (inhaled short- or long-acting beta-agonists, inhaled corticosteroids, or short- or long-acting anticholinergics) for 28 weeks in Periods IV and V (EXT2)
Arm/Group | MK-0873 0.75 mg Base Study | MK-0873 1.25 mg Base Study | MK-0873 2.5 mg Base Study | Placebo Base Study | MK-0873 2.5 mg EXT 1 | Placebo EXT 1 | MK-0873 2.5 mg + Usual Care EXT 2 | Usual Care EXT2
Serious Adverse Events (participants affected / at risk) | 10/150 | 11/148 | 10/153 | 6/153 | 17/317 | 4/107 | 9/187 | 5/71
Other Adverse Events (participants affected / at risk) | 47/150 | 42/148 | 66/153 | 43/153 | 72/317 | 19/107 | 37/187 | 11/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0873 0.75 mg Base Study (N=150) | MK-0873 1.25 mg Base Study (N=148) | MK-0873 2.5 mg Base Study (N=153) | Placebo Base Study (N=153) | MK-0873 2.5 mg EXT 1 (N=317) | Placebo EXT 1 (N=107) | MK-0873 2.5 mg + Usual Care EXT 2 (N=187) | Usual Care EXT2 (N=71)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 4 (4) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 6 (6) | 2 (3) | 3 (3) | 2 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0873 0.75 mg Base Study (N=150) | MK-0873 1.25 mg Base Study (N=148) | MK-0873 2.5 mg Base Study (N=153) | Placebo Base Study (N=153) | MK-0873 2.5 mg EXT 1 (N=317) | Placebo EXT 1 (N=107) | MK-0873 2.5 mg + Usual Care EXT 2 (N=187) | Usual Care EXT2 (N=71)
Diarrhoea (Gastrointestinal disorders) | 12 (15) | 7 (9) | 20 (29) | 3 (3) | 16 (17) | 3 (5) | 8 (9) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 9 (9) | 3 (3) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (13) | 14 (21) | 19 (22) | 13 (16) | 18 (22) | 4 (4) | 16 (21) | 4 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 29 (34) | 26 (30) | 32 (42) | 28 (35) | 40 (52) | 13 (15) | 18 (21) | 7 (8)

LIMITATIONS AND CAVEATS:
The extension studies were terminated based on data from the completed base study suggesting that MK-0873, at doses up to 2.5 mg per day, demonstrated no benefits versus placebo in lung function or symptoms in participants with COPD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.